CLINICAL TRIAL: NCT01581528
Title: Metabolic Pathways in T-Cell Acute Lymphoblastic Leukemia (T-ALL)
Brief Title: Studying Samples From Patients With T-Cell Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL12B5; COG-AALL12B5 (Other: clinicaltrials.gov); AALL12B5 (Other: Children's Oncology Group); NCI-2012-00728 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: T-cell childhood acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; T-cell adult acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Gene Expression Profiling; Cell Culture Techniques; Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Other: cell culture procedure
Other: flow cytometry
Other: laboratory biomarker analysis
Other: metabolic assessment

SUMMARY:
RATIONALE: Studying samples of blood, tissue, and bone marrow from patients with cancer in the laboratory may help doctors identify learn more about biomarkers related to cancer. It may also help doctors to find better ways to treat cancer.

PURPOSE: This research studies samples from patients with T-cell acute lymphoblastic leukemia (T-ALL).

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the metabolic status and regulation of primary T-cell acute lymphoblastic leukemia (T-ALL) relative to control resting peripheral T cells.
* Establish the effects of metabolic inhibition on metabolic stress pathways and apoptosis.
* Determine how metabolic inhibition interacts with chemotherapy or targeted therapy drugs to kill T-ALL cells.

OUTLINE: T-ALL samples cultured alone or with gamma secretase inhibitors (GSI) or PI3K inhibitors are analyzed for metabolic characteristics including glucose transporter 1 (Glut1) expression, mitochondrial mass, phospho-flow for 5' adenosine monophosphate-activated protein kinase (AMPK), acetyl-CoA carboxylase (ACC), and mammalian target of rapamycin (mTOR) by flow cytometry. T-ALL samples and normal CD4+ T cells (control) are also exposed to ± 2-deoxyglucose or ± the glutaminolysis inhibitor media and analyzed for metabolic stress responses over time in particular, AMPK activation, autophagy (immunofluorescence for LC3-II processing), and BCL2-associated X protein (Bak) and Bax activation to indicate apoptosis. These cells (T-ALL and control) are then cultured with cyclophosphamide, dexamethasone, or the B-cell CLL/lymphoma 2 (Bcl-2) inhibitor, ABT-737, to determine cell death over time.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Sample from patients diagnosed with T-ALL
* Samples from independent healthy donors obtained through the Gulf Coast Regional Blood Center (controls)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with T-ALL
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Metabolic status of primary T-ALL
Effects of metabolic inhibition on metabolic stress pathways and apoptosis
Metabolic inhibition interaction with chemotherapy or targeted drugs

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey C. Rathmell, PhD, Principal Investigator — Duke Cancer Institute